CLINICAL TRIAL: NCT03313557
Title: An Open-label, Non-randomised, Multicentre Study to Allow Continued Access to and Assess the Safety and Tolerability of AZD1775 for Patients Enrolled in AZD1775 Clinical Pharmacology Studies
Brief Title: AZD1775 Continued Access Study to Assess Safety and Tolerability for Patients Enrolled in AZD1775 Clinical Pharmacology Studies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D6014C00007
Record Dates: First submitted 2017-10-13; First posted 2017-10-18 (Actual); Last update posted 2019-06-24 (Actual); Status verified 2019-06

CONDITIONS: Solid Tumors
Keywords: Continued access, safety assessments

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Wee-1 kinase inhibitor AZD1775 (Experimental): To assess the safety of AZD1775 following oral dosing of the capsule formulation in patients with advanced solid tumours in patients who have previously completed 1 of the AZD1775 clinical pharmacology studies and not have met any requirements to permanently discontinue treatment with AZD1775.
  Interventions: Drug: Wee-1 kinase inhibitor AZD1775

INTERVENTIONS:
Drug: Wee-1 kinase inhibitor AZD1775 — Patients will receive AZD1775 300 mg orally once daily. Days 1 to 5 and 8 to 12 of a 21 day cycle (ie, 5 days on and 2 days off for Weeks 1 and 2 of a 21-day cycle). All patients must receive a serotonin receptor 3 (5-HT3) antagonist, ondansetron (Zofran) 8 mg orally/IV or granisetron (Kytril) 1 mg orally/IV prior to each dose of AZD1775. Dexamethasone 4 mg orally/IV will be given with each AZD1775 dose at a minimum on the first day of dosing of AZD1775 of every 5 day dosing period, unless contraindicated or not well-tolerated.

SUMMARY:
Open-label, non-randomised study to provide continued access to AZD1775 for patients with advanced solid tumours who have previously completed an AZD1775 clinical pharmacology study and to investigate the safety of AZD1775.

DETAILED DESCRIPTION:
This is an open-label, non-randomised study designed to provide continued access to AZD1775 for eligible patients with advanced solid tumours who have previously completed an AZD1775 clinical pharmacology study and to investigate the safety of a once daily monotherapy regimen of AZD1775 in patients with advanced solid tumours.

All patients who completed 1 of the parent clinical pharmacology studies are eligible for this study after a washout period of at least 4 days (minimum duration defined in the parent study protocol) and meet the eligibility criteria specified in this protocol. Patients who discontinue early from the parent study will be considered by the Sponsor and treating physician on a case-by-case basis.

During the study, patients will continue to receive AZD1775 as long as they are benefiting from treatment in the Investigator's opinion and do not meet any other discontinuation criteria.

ELIGIBILITY:
Inclusion Criteria:

For inclusion in this study, patients must fulfil the following criteria:

* Has read and understands the informed consent form (ICF) and has given written informed consent prior to any study procedures.
* Female or male aged ≥18 years.
* Has completed 1 of the parent AZD1775 clinical pharmacology studies (ie, D6014C00002, D6014C00003, D6014C00004, D6014C00005, or D6014C00006) and in the Investigator's opinion will continue to benefit from treatment with AZD1775. Patients who discontinue early from the parent study will be considered by the Sponsor and treating physician on a case-by-case basis.
* Any prior radiation must have been completed at least 7 days prior to the start of study treatment, and patients must have recovered from any acute effects prior to the start of study treatment.
* Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 to 1.
* Baseline laboratory values within 7 days of study treatment initiation in the CA study:

  * Absolute neutrophil count (ANC) ≥1500/μL.
  * Haemoglobin ≥9 g/dL.
  * Platelets ≥100,000/μL.
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3 x upper limit of normal (ULN) or ≤5 x ULN if known hepatic metastases.
  * Serum bilirubin within normal limits or ≤1.5 x ULN in patients with liver metastases; or total bilirubin ≤3.0 x ULN with direct bilirubin within normal limits in patients with well documented Gilbert's Syndrome.
  * Serum creatinine ≤1.5 x ULN, or measured creatinine clearance (CrCl) calculated by Cockcroft-Gault method ≥45 mL/min (confirmation of creatinine clearance is only required when creatinine is >1.5 x ULN) CrCl (glomerular filtration rate) = (140-age) x (weight/kg) x Fa (72 x serum creatinine mg/dL) where F = 0.85 for females and F = 1 for males.
* Female patients who are of non-childbearing potential and fertile women of childbearing potential (WoCBP) who agree to use adequate contraceptive measures that are in place during screening (or consent), for the duration of the study, and for 1 month after treatment stops; who are not breastfeeding; and who have a negative serum or urine pregnancy test prior to the start of study treatment.
* Male patients must be willing to use barrier contraception (ie, condoms) for the duration of the study and for 3 months after study treatment discontinuation.
* Willingness and ability to comply with the study and the follow-up procedures.

Exclusion Criteria:

Patients must not enrol in this study if any of the following exclusion criteria are fulfilled:

* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca personnel and/or personnel at the study centre).
* Previous enrolment and received study treatment in the present study. Patients can, however, be re-screened if the reason for the screen failure no longer exists.
* Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or the follow-up period of an interventional study.
* Must not have received another systemic anti-cancer therapy in the interval following participation in the AZD1775 clinical pharmacology study and the start of treatment on the CA protocol.
* Not developed any clinical findings suggestive of brain metastasis. Patients continue to be neurological stable and remain off systemic corticosteroids following treatment of known brain metastases.
* Did not tolerate AZD1775 in the parent study in the opinion of the Investigator.
* Where a course of palliative radiotherapy was indicated, the last fraction must have been delivered before the start of study treatment on the CA study.
* Major surgical procedures ≤28 days of beginning study treatment, or minor surgical procedures ≤7 days. No waiting period required following port-a-cath placement or other central venous access placement.
* Grade >1 toxicities from prior therapy, according to the Common Terminology Criteria for Adverse Events (CTCAE), excluding alopecia or anorexia.
* Continue to be able to swallow oral medication, did not undergo placement of a percutaneous endoscopic gastrostomy tube and did not require total parenteral nutrition.
* Has had prescription or non-prescription drugs or other products known to be sensitive to CYP3A4 substrates or CYP3A4 substrates with a narrow therapeutic index, or to be moderate to strong inhibitors/inducers of CYP3A4 between the parent study and entry into this CA study. Co administration of aprepitant or fosaprepitant during this study is prohibited.
* Has consumed herbal preparations between the parent study and entry into this CA study.
* Has consumed grapefruit, grapefruit juice, Seville oranges, Seville orange marmalade, or other products containing grapefruit or Seville oranges between the parent study and entry into the CA study.
* Any known hypersensitivity or contraindication to AZD1775 or to the components thereof.
* Any of the following cardiac diseases currently or within the last 6 months as defined by the New York Heart Association ≥Class 2:

  * Unstable angina pectoris.
  * Congestive heart failure.
  * Acute myocardial infarction.
  * Conduction abnormality not controlled with pacemaker or medication.
  * Significant ventricular or supraventricular arrhythmias (patients with chronic rate-controlled atrial fibrillation in the absence of other cardiac abnormalities are eligible).
* AZD1775 should not be given to patients who have a history of Torsades de pointes unless all risk factors that contributed to Torsades have been corrected. AZD1775 has not been studied in patients with ventricular arrhythmias or recent myocardial infarction.
* Patient with mean resting QTc interval (specifically QTc calculated using the Fridericia formula [QTcF]) >450 ms for males and >470 ms for females from 3 electrocardiograms (ECGs) performed within 2 to 5 minutes apart during screening, or congenital long QT syndrome.
* Pregnant or lactating female patients.
* Serious, symptomatic active infection at the time of study entry, or another serious underlying medical condition that would impair the ability of the patient to receive study treatment.
* Active infection with hepatitis B, hepatitis C, or human immunodeficiency virus (HIV).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-10-27 (Actual); Primary Completion 2019-05-17 (Actual); Study Completion 2019-05-17 (Actual)

PRIMARY OUTCOMES:
Adverse Events, graded by the National Cancer Institute Common Terminology Criteria for Adverse Event's (CTCAE v4.3) | Until 30 days following the final dose of AZD1775
  To assess the safety of AZD1775 following oral dosing of the capsule formulation in patients with advanced solid tumours
Complete physical examination including performance status assessed using the Eastern Cooperative Oncology Group (ECOG) Performance Status criteria. | Until 30 days following the final dose of AZD1775
  To assess the safety and tolerability of AZD1775 printed capsules following oral dosing in patients with advanced solid tumours. If new or aggravated physical findings imply deterioration compared with baseline, the finding will be reported as an Adverse Event, unless the findings are unequivocally due to disease progression.
Pulse Rate (beats/min) | Until 30 days following the final dose of AZD1775
  To assess the safety and tolerability of AZD1775 printed capsules following oral dosing in patients with advanced solid tumours.
Blood Pressure (mm Hg) | Until 30 days following the final dose of AZD1775
  To assess the safety and tolerability of AZD1775 printed capsules following oral dosing in patients with advanced solid tumours.
Body Temperature (°C) | Until 30 days following the final dose of AZD1775
  To assess the safety and tolerability of AZD1775 printed capsules following oral dosing in patients with advanced solid tumours.
Evaluation of Laboratory Parameters | Until 30 days following the final dose of AZD1775
  To assess the safety and tolerability of AZD1775 printed capsules following oral dosing in patients with advanced solid tumours; deterioration of haematology and clinical chemistry laboratory values as compared to baseline will be reported as Adverse Events if they fulfill any of the Serious Adverse Events criteria or are the reason for discontinuation of the study treatment unless clearly due to the progression of disease under study; if deterioration in a laboratory value is associated with clinical signs and symptoms, the sign or symptom will be reported as an AE and the associated laboratory result will be considered as additional information.

CONTACTS AND LOCATIONS:
Overall Officials: Lone Ottesen, MD, Study Director — AstraZeneca; Henk Verheul, MD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (13):
- United States (7):
  - Research Site, Bingham Farms, Michigan
  - Research Site, Detroit, Michigan
  - Research Site, Lebanon, New Hampshire
  - Research Site, Cincinnati, Ohio
  - Research Site, Providence, Rhode Island
  - Research Site, Greenville, South Carolina
  - Research Site, Dallas, Texas
- France (2):
  - Research Site, Bordeaux
  - Research Site, Saint-Herblain
- Netherlands (2):
  - Research Site, Amsterdam
  - Research Site, Maastricht
- United Kingdom (2):
  - Research Site, Glasgow
  - Research Site, Manchester

IPD SHARING:
Plan to Share IPD: No